CLINICAL TRIAL: NCT03879616
Title: Optimizing the Use of Reminders for Gastrointestinal Procedure Appointments
Brief Title: Optimizing Gastrointestinal Procedure Appointments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GI2019
Record Dates: First submitted 2019-03-08; First posted 2019-03-19 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Gastrointestinal Disease
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An Enhanced Reminder (Experimental): Members randomized to this arm of the study will receive an enhanced reminder protocol, which will include multiple reminders, multiple modalities, and motivational messages. The timing of reminders will depend on the wait time between the date the appointment is made and the date of the appointment.
  * An email reminder will be sent to all members who have provided their personal email information.
  * Members will receive up to two text messages that "roll over" to an IVR automated phone call if the text cannot be delivered.
  * Members scheduled for colonoscopy will also receive a single IVR-T reminder to begin their bowel prep the morning of the calendar day prior to the procedure.
  Interventions: Behavioral: An Enhanced Reminder
- Control (Other): Members randomized to this arm of the study will receive a single text message that "rolls over" to an IVR automated phone call if the text cannot be delivered. This message will be delivered 7 business days prior to the appointment. This replicates the current protocol for GI procedures. Of note, members who schedule appointments within 7 days of the procedure currently receive no reminders.
  Interventions: Behavioral: An Enhanced Reminder

INTERVENTIONS:
Behavioral: An Enhanced Reminder — This study will be a randomized trial over a 6-month period (March 8 through September 7, 2019) in 3 GI endoscopy clinics (Franklin, Rock Creek, and Lone Tree). All members currently receive a text reminder 7 days prior to their procedure, which rolls over to a telephone reminder if the text cannot be delivered or the member's phone is not text-enabled. Members will be randomized either to receive this standard IVR-T protocol (control) or to receive an enhanced reminder (intervention) protocol.
  Data from the randomized trial, for both intervention and control participants, will be analyzed to develop a statistical prediction rule that identifies members at highest risk of missing their procedure.

SUMMARY:
This project will address the question:

Does an "enhanced" IVR-T protocol differ in effectiveness from the standard IVR-T protocol in reducing missed appointments and late cancellations for GI endoscopy? Hypothesis: The enhanced IVR-T protocol will be more effective.

DETAILED DESCRIPTION:
This study will be a randomized trial over a 6-month period (March 8 through September 7, 2019) in 3 GI endoscopy clinics (Franklin, Rock Creek, and Lone Tree). All members currently receive a text reminder 7 days prior to their procedure, which rolls over to a telephone reminder if the text cannot be delivered or the member's phone is not text-enabled. Members will be randomized either to receive this standard IVR-T protocol (control) or to receive an enhanced reminder (intervention) protocol.

Randomization: Beginning in March 8, 2019, a randomization algorithm will be used in the Structured Query Language program that manages the IVR relational database to assign each visit for a procedure at all three sites to control or intervention. Since members with multiple procedures on different days during the study period could receive control or intervention for different visits, the statistical analysis will be limited to the first randomized appointment during the project period. Randomization will be stratified by clinic site.

ELIGIBILITY:
Inclusion criteria:

* Members scheduled for any GI procedure (upper endoscopy, colonoscopy, or both), with or without anesthesia, at all three clinical sites (Franklin, Rock Creek, Lone Tree) will be included if their procedure is scheduled ≥ 2 days prior to the procedure. The IVR-T protocol will be adapted based on the wait time between appointment scheduling and the date of the procedure.
* Members with all clinical indications (screening, diagnosis, or surveillance), will be included.

Exclusion criteria:

* KPCO members who request not to participate in research or not to receive IVR-T or email outreach
* KPCO members in the "break the glass" or "code pink" protocols.
* Members whose procedure is scheduled < 2 days prior to the procedure.

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15974 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-09-08 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Cancellation and Rate of Missed Appointments | 6 months
  The primary outcome for the study will be "appointment loss," defined by GI leaders as the combined rate of prior day cancellations, same-day cancellations, and missed clinic appointments ("no shows"). The rationale for this outcome definition is that it is difficult to schedule new procedures within this time frame.

SECONDARY OUTCOMES:
The Boston Bowel Preparation Measure | 6 months
  A secondary outcome will be the assessment of the adequacy of the bowel preparation for colonoscopy only.

CONTACTS AND LOCATIONS:
Overall Officials: John Steiner, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT03879616/Prot_SAP_000.pdf